CLINICAL TRIAL: NCT05277519
Title: Neuroplasticity Induced by Functional Muscle Tendon Vibrations in Patients With Acquired Brain Injury
Brief Title: Neuroplasticity After Proprioceptive Rehabiliation
Acronym: VibraLCA
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-11; 2021-A00822-39 (Registry Identifier: ID RCB)
Record Dates: First submitted 2021-09-16; First posted 2022-03-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Hemiparesis; Traumatic Brain Injury
Keywords: Neuroplasticity; Electrophysiology; MRI; Neurophysiology; Muscle vibration
MeSH Terms: conditions — Stroke; Paresis; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vibrations — Sequenced muscle vibrations during 30 min., 3 times a week during 5 weeks

SUMMARY:
Sequences of muscle tendon vibrations allow to reproduce the sensory feedback during movement like locomotion and kinaesthesia. It is known that such a treatment promotes motor recovery after stroke assuming that it enhances neuroplasticity. The aim of the research is to study the activity in cerebrospinal circuitry to evaluate the neuroplastic changes during and after instrumented proprioceptive rehabilitation relying on sequences of muscle vibration in subacute stroke stages.

DETAILED DESCRIPTION:
Randomized control trial : 28 patients with active vibrations vs. 28 patients with sham stimulation Subacute phase : D15 to 6 months after stroke or patients with traumatic brain injury with similar semiology as stroke (hemiparesis) Measure at baseline : Electrophysiological investigations (EMG,EEG, MRI, clinical evaluation) Treatment of 5 weeks with 3 sessions of vibrations or sham a week Evaluation at mid time (electrophysiology and clinical examinations) Final examination (electrophysiology, MRI and clinical examination)

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis at least transient in lower limb following an acquired brain injury (stroke or traumatic brain injury)
* French spoken
* Affiliated to a French social insurance
* No previous traumatic, vascular or neurodegenerative injuries
* Having presented during the acute phase or presenting a motor deficit of one of the lower limbs
* Presenting an absence of autonomy of walking at the entrance of the rehabilitation department
* In the sub-acute phase, i.e. from 15 days to 6 months after the accident
* Presenting moderate cognitive disorders allowing them to understand instructions and give their consent

Exclusion Criteria:

* strong cognitive disorders
* maintenance of justice, tutelage, legal guardianship
* Pregnancy and breastfeeding
* Outpatients who do not have weekly follow-up in the rehabilitation department

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 56 patients randomly affected to the experimental group receiving active vibration or sham
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Baseline EMG | Evaluation at baseline (4 days before treatment)
  H-reflex and reciprocal inhibition
Baseline EEG | Evaluation at baseline (4 days before treatment)
  SEP and resting state activity
EMG change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  H-reflex and reciprocal inhibition
EEG change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  SEP and resting state activity
EMG change after the 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  H-reflex and reciprocal inhibition
EEG change after the 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  SEP and resting state activity

SECONDARY OUTCOMES:
Baseline MD | Evaluation at baseline (4 days before treatment)
  Evaluation of white matter integrity along the corticospinal tract by calculating the mean diffusivity (MD) evaluated from diffusion MRI
Baseline FA | Evaluation at baseline (4 days before treatment)
  Evaluation of white matter integrity along the corticospinal tract by calculating the fraction of anisotropy (FA) evaluated from diffusion MRI
Baseline Muscle Strength | Evaluation at baseline (4 days before treatment)
  score to Medical Research Council scale
Muscle Strength change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  score to Medical Research Council scale
Muscle Strength change from baseline after 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  score to Medical Research Council scale
Baseline Spasticity | Evaluation at baseline (4 days before treatment)
  score to Modified Ashworth scale
Spasticity change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  score to Modified Ashworth scale
Spasticity change from baseline after 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  score to Modified Ashworth scale
Baseline sensorimotor function | Evaluation at baseline (4 days before treatment)
  subscore for lower limbs to Fugl meyer assessment
Sensorimotor function change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  subscore for lower limbs to Fugl meyer assessment
Sensorimotor function change from baseline after 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  subscore for lower limbs to Fugl meyer assessment
Baseline Balance | Evaluation at baseline (4 days before treatment)
  Score to Berg balance scale
Balance change from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  Score to Berg balance scale
Balance change from baseline after 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  Score to Berg balance scale
Baseline walking | Evaluation at baseline (4 days before treatment)
  score to 10-m walking test
Walking from baseline after 2-week treatment | Evaluation during the 3rd week of treatment
  score to 10-m walking test
Walking from baseline after 5-week treatment | Evaluation 4 days after the end of the 5-week treatment
  score to 10-m walking test
Change in MD | Evaluation 4 days after the end of the 5-week treatment
  Evaluation of white matter integrity along the corticospinal tract by calculating the mean diffusivity (MD) evaluated from diffusion MRI
Change in FA | Evaluation 4 days after the end of the 5-week treatment
  Evaluation of white matter integrity along the corticospinal tract by calculating the fraction of anisotropy (FA) evaluated from diffusion MRI

CONTACTS AND LOCATIONS:
Overall Officials: Eleonore Bayen, MD, PhD, Principal Investigator — Sorbonne University - AP-HP (Pitié-Salpêtrière Hospital)
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided